CLINICAL TRIAL: NCT03971045
Title: Combination of Pembrolizumab With Oral Metronomic Cyclophosphamide in Patients With Chest Wall Breast Cancer (PERICLES): A Phase II Study
Brief Title: Pembrolizumab and Oral Metronomic Cyclophosphamide in Patients With Chest Wall Breast Cancer
Acronym: PERICLES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 675
Record Dates: First submitted 2019-05-20; First posted 2019-06-03 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Chest Wall Tumor
Keywords: Pembrolizumab; Immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Phase II single center, open-label, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab and metronomic cyclophosphamide (Experimental): .Patients will be treated with pembrolizumab administered as an intravenous infusion at 200 mg in 21-day treatment cycles and oral cyclophosphamide (CTX) 50 mg per day in metronomic administration as a 21 days cycle
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Patients will be treated with pembrolizumab administered as an intravenous infusion at 200 mg in 21-day treatment cycles and oral cyclophosphamide (CTX) 50 mg per day in metronomic administration as a 21 days cycle
  Other Names: Cyclophosphamide

SUMMARY:
This is a Phase II single center, open-label, non-randomized study in patients with locally recurrent, inoperable, and/or metastatic inflammatory breast cancer with lymphangitic spread to the chest wall. Patients will be treated with pembrolizumab administered as an intravenous infusion at 200 mg in 21-day treatment cycles and oral cyclophosphamide (CTX) 50 mg per day in metronomic administration as a 21 days cycle Forty-six patients will be required for the study. Key inclusion criteria are PDL1 (≥1%) positive and/or tumor infiltrating lymphocyte positive (≥1%) locally advanced "chest wall" breast cancer (with or without distant metastases), who have been treated with chemotherapy or radiation therapy may be eligible for this study. Patients with cutaneous metastases only (with or without evidence of primary tumor) are eligible for the study. Key exclusion criteria included prior anti PD1 or anti CTLA-4 or other immune pathway-targeted therapy. Patients with autoimmune diseases and/or receiving drugs who interfere with the immune system will not be eligible.

DETAILED DESCRIPTION:
This is a Phase II single center, open-label, non-randomized study in patients with locally recurrent, inoperable, and/or metastatic inflammatory breast cancer with lymphangitic spread to the chest wall. Patients will be treated with pembrolizumab administered as an intravenous infusion at 200 mg in 21-day treatment cycles and oral cyclophosphamide (CTX) 50 mg per day in metronomic administration as a 21 days cycle. Forty-six patients will be required for the study. The study will be open to participants with histologically confirmed, inoperable, locally recurrent and/or metastatic breast cancer (mBC) with lymphangitic spread to the chest wall (chest wall disease), which had received one or more prior cytotoxic treatment. Key exclusion criteria consist of prior anti-PD1, anti-CTLA-4 or other immune pathway-targeted therapy. Patients with autoimmune diseases and/or receiving drugs who interfere with the immune system will not be eligible. Patients will be monitored carefully for the development of adverse experiences and will be monitored for clinical and/or radiographic evidence of disease progression according to usual standards of clinical practice. Adverse experiences will be evaluated according to criteria outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. For individual patients that experience dose-limiting toxicities, criteria for dose modification of pembrolizumab and CTX are outlined in details in the protocol. Treatment with pembrolizumab and metronomic chemotherapy will continue until documented disease progression, unacceptable adverse events (as reported by the site), intercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, completion of 24 months of treatment with pembrolizumab, or administrative reasons requiring the cessation of treatment. Subjects who attain complete response (CR) confirmed by central radiology review may consider stopping trial treatment after receiving at least 24 weeks of treatment. Subjects who discontinue treatment after 24 months of therapy for reasons other than disease progression or intolerability or who discontinue treatment after attaining a CR may be eligible for up to one year of retreatment after they have experienced radiographic disease progression. The decision to retreat will be at the discretion of the Investigator, only if no cancer treatment was administered since the last dose of pembrolizumab, the subject still meets the safety parameters listed in the Inclusion/Exclusion criteria and the trial remains open.

Primary Objective: assessment of the efficacy of pembrolizumab and metronomic cyclophosphamide according to immune-related RECIST (irRECIST) criteria in patients with chest wall breast cancer. Primary endpoint will be objective response (confirmed CR or PR as best overall response) based on irRECIST criteria and also based on evaluable disease.

Secondary objectives: duration of response (DoR); time to progression (TTP); progression-free survival (PFS); overall survival (OS).

Exploratory Objectives: responses according to levels of PD-L1, measured by immunohistochemistry IHC in unresectable locoregional lesion. Responses according to levels of tumor infiltrating lymphocytes. Responses according to ER status. Responses according to FISH ratio and HER2 copy number. Tumor dynamics during the disease course as well as emergence of new clones (i.e.: resistance mechanisms) by determination of circulating tumor DNA (ctDNA). Sequencing of material from tumor biopsies to determine molecular profiles of responders and non-responders. Evaluation of efficacy by immune-related RECIST (irRECIST) (i.e.: irORR, irDoR, irPFS, irDCR). Through analysis of peripheral blood transcriptome in patients treated with pembrolizumab and cyclophosphamide therapy (P and CTX) combination therapy the investigators aim at:

1. Defining baseline peripheral blood gene signatures associated with treatment responsiveness (pre-treatment biomarkers);
2. Defining molecular perturbations associated with the administration P and CTX combination therapy and their relationship with immune-related adverse events (post-treatment predictive biomarkers) and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, PDL1 (≥1%) positive and/or tumor infiltrating lymphocytes (TILs) positive (≥1%), locally advanced "chest wall" breast cancer (with or without distant metastases), who have been treated with chemotherapy or radiation therapy may be eligible for this study. Patients with cutaneous metastases only (with or without evidence of primary tumor) are also eligible;
* Patients must have tissue accessible for serial biopsies;
* Expected survival of > 3 months;
* Be willing and able to provide written informed consent/assent for the trial. The subject may also provide consent/assent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor;
* Be 18 years of age on day of signing informed consent;
* Be a female or male subject with IBC with lymphangitic spread to the chest wall. ER, PgR and HER2 status determination is required for enrollment;
* Have provided tissue for PD-L1 biomarker analysis from a newly obtained core or excisional biopsy of a tumor lesion (mandatory) and received permission for enrollment from the Core Lab based on the adequacy of the biopsy specimen. Repeat samples may be required if adequate tissue is not provided;
* Have measurable metastatic disease based on irRECIST criteria as determined by central radiology review. Tumor lesions situated in a previously irradiated area are considered measurable, if progression has been demonstrated in such lesions. Note: The exact same image acquisition and processing parameters should be used throughout the study;
* Have a performance status of 0 or 1 on the ECOG Performance Scale. Assessment should be performed within 10 days of treatment initiation;
* Female subjects of childbearing potential (Section 2.9.2) must be willing to use an adequate method of contraception as outlined in Section 2.9.2 - Contraception, for the course of the study through 120 days after the last dose of study medication;
* Male subjects childbearing potential (Section 2.9.2) must agree to use an adequate method of contraception as outlined in Section 2.9.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject;
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
* Patients with hormone receptor-positive and/or HER2-positive breast cancer would be eligible for the study only if their disease is considered refractory to hormonal or anti-HER2 agents, respectively, and no further hormonal or anti-HER2 treatment is indicated;
* Demonstrate adequate organ function as defined in protocol, all screening labs should be performed within 10 days of treatment initiation;
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
* Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject;
* Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment;
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment;
* Has a known history of active TB (Bacillus Tuberculosis);
* Hypersensitivity to pembrolizumab or any of its excipients;
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier;
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note 1: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note 2: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer;
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment;
* Has known history of, or any evidence of active, non-infectious pneumonitis;
* Has an active infection requiring systemic therapy;
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator;
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment;
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent;
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies);
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response | Participants will be followed for the duration of treatment, an expected average of 6-months
  Confirmed CR or PR as best overall response based on irRECIST criteria

SECONDARY OUTCOMES:
Duration of response (DoR) | Participants will be followed for the duration of treatment, an expected average of 6-months
  In months
Progression-free survival (PFS) | Progression-free survival assessed at 24 months
  In months
Overall survival (OS) | Overall survival assessed up to 24 months
  In months

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data will de decided if opportunity of collaborations will emerge
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code